# STUDY PROTOCOL

Protocol Title The Effect of Enstilar versus Vehicle on Target Lesions

in Moderate Plaque Type Psoriasis Patients

Protocol Date March 20, 2018

Protocol # ENS-1702

Investigator/Sponsor Leon Kircik, MD Skin Sciences, PLLC

1169 Eastern Parkway, Suite 2310

Louisville, KY 40217

## **PROTOCOL SIGNATURE PAGE**

The signature below constitutes the approval of this protocol and the supplements, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality. This study will be conducted per protocol according to local legal and regulatory requirements, and in accord with the spirit of GCP. However, will not adhere to the requirements of the comprehensive ICH-GCP guidelines.

| Investigator | | |
|--------------|-----------|------|
| Printed Name | Signature | Date |

## 1 STUDY OBJECTIVE

#### 2 STUDY DESIGN

This will be a 3-center, open label study. 24 subjects will be enrolled. Target lesion will be identified on either the knees or elbows and evaluated for efficacy (TLSS) for the secondary endpoints at baseline, week 2 and week 4 (secondary). PGA will be recorded at baseline, week 2 and week 4 (primary endpoint). TLSS is expected to be a minimum score of 2 (moderate) for erythema, 2 (moderate) scaling, 2 (moderate) plaque thickness with overall score of 6. The study will consist of screening/baseline, week 2 & week 4. (3 visits). Adverse events will be recorded throughout study. Selected patient target lesions will be photographed at baseline, week 2 & week 4. Patients will be instructed to apply a 2 sec spray time per 1% BSA on plaques and instructed to wash their hands thoroughly after application.

Subjects will attend a Screening Visit/Baseline visit and if found eligible will be randomized to study treatment. Patients will be counselled on the use of the study medication and the medications will be labelled for the appropriate group as noted above. The duration of the study is 4 weeks and consists of a Screening/Baseline visit, and one (1) Follow-up Visit at Week 2 and end of treatment visit at week 4.

## 3 SELECTION AND WITHDRAWAL OF SUBJECTS

#### 3.1 Inclusion Criteria

## Inclusion:

i. 1. Outpatient, male or female subjects of any race, 18 years of age or higher. Female subjects of childbearing potential must have a (-)UPT result at within 7 days of the first dose of study drug and practice a reliable method of contraception throughout the study;

A female is considered of childbearing potential unless she is:

- postmenopausal > 5Y, without a uterus and/or both ovaries; or has been surgically sterile for > 6M.

Reliable methods of contraception are:

- hormonal methods or IUD in use > 90d prior to study drug administration, barrier methods plus spermicide in use > 14d prior, or vasectomized partner.

[Exception: Female subjects of CBP who are not sexually active are not required to practice a reliable method of contraception and may be enrolled at the Investigator's discretion provided they are counselled to remain sexually inactive for the duration of the study and understand the risks involved in getting pregnant during the study.

- ii. Moderate plaque type psoriasis eligible for topical therapies.
- iii. Patients with a minimum of 3% BSA to a maximum of 20% BSA & bilateral symmetric psoriatic plaques of 2 to 4 cm in diameter
- iv. Physician Global Assessment (PGA) score of 3.
- v. Able to understand study requirements and sign Informed Consent/HIPAA forms.

#### **Exclusion:**

- i. Female subjects who are pregnant, breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control, or male subjects planning a pregnancy with their spouse or partner while in the study.
- ii. History of hypercalcaemia or vitamin D toxicity.
- iii. Patients with guttate, erythrodermic, or pustular psoriasis
- iv. Serious skin condition (other than psoriasis) or uncontrolled medical condition (in the opinion of the investigator).
- v. Topical steroids, topical immunomodulators, topical vitamin D derivatives, tar, salicylic acid, anthralin or any other topical treatment for psoriasis within 2 weeks of baseline.
- vi. Use of any biologics within 3 months of baseline.
- vii. Use of other systemic psoriasis treatments (ie, oral retinoids, methotrexate, cyclosporine, or other immunomodulators) within 4 weeks of baseline.
- viii. Use of UVB or PUVA within 2 weeks of baseline.
- ix. Skin conditions (e.g. eczema) psoriasis that may interfere with evaluations of psoriasis.
- x. Known hypersensitivity to Enstilar or any of its components.
- xi. Contraindications according to Enstilar
- xii. Current drug or alcohol abuse (Investigator opinion).
- xiii. Subject unable to commit to all the assessments required by the protocol

## 3.3 Withdrawal of Subjects

It is the right and duty of the Investigator to discontinue the study participation of a subject when the subject's health or well-being is threatened by continuation in the study. Such subjects should be withdrawn from the study and not continued under a modified regimen. The following are circumstances that would result in the subject's discontinuation from the study:

- the subject experiences a serious adverse event rendering them unable to continue study participation;
- the subject is unable to physically or mentally tolerate the use of the test medication;
- an exclusion criterion becomes apparent at any time during the study; or
- the subject voluntarily withdraws.

In the event of premature discontinuation from the study, the Investigator should determine the primary reason for discontinuation.

If a subject withdraws for any reason, the subject will be replaced.

## 4 TREATMENT OF SUBJECTS AND FOLLOW-UP

# 4.1 Study Procedures

# 4.1.1 Assessment Schedule

| Procedures/Non-Procedure Description | Screening<br>and<br>Baseline | Week 2 | Week 4 |
|---|---|---|---|
| Informed Consent | Х | | |
| Medical History and Demographics | Х | | |
| Inclusion/Exclusion Criteria | Х | | |
| Initial Prior/Concurrent Medications | X | | |
| Concurrent Medications subsequent visit | X | Х | X |
| Vital Signs (includes height/weight for initial visit only) | Х | Х | X |
| Complete Physical Examination | X | | Х |
| TLSS scoring | X | Х | X |
| Pregnancy Test (female subject of childbearing potential only) | X | | Х |
| Photography of Target Lesion<br>(investigator will supply all<br>photographic equipment and<br>background) * | X | X | X |
| Adverse event assessment and reporting if applicable | Х | Х | X |
| Clinical severity/efficacy<br>assessments by investigator (BSA,<br>PGA) | X | Х | X |
| Pharmacy Dispense/Drug Accountability | Х | Х | Х |

<sup>\*</sup>At select sites only

# 4.1.2 Screening Visit/ Baseline Visit

- Informed Consent/HIPAA
- Urine Pregnancy Test (if applicable)
- Subject Demographics/Medical History
- Concomitant Medication/Treatment
- Inclusion/Exclusion Criteria
- Assessments

- BSA (Affected Body Surface Area)
- PGA
- Identification of target lesion
- Photography of target lesion at select sites only
- TLSS
- Physical Exam
- Vital Signs / Height & Weight
- Drug dispensation
- Adverse events
- Cutaneous adverse events

## Week 2

- Concomitant Medication/Treatment
- Assessments
  - BSA (Affected Body Surface Area)
  - PGA
  - Photography of target lesion at select sites only
  - TLSS
- Vital Signs
- Drug dispensation
- Adverse events
- Cutaneous adverse events

#### 4.1.3 Week 4/End of treatment

- Concomitant Medication/Treatment
- Assessments
  - BSA (Affected Body Surface Area)
  - PGA
  - Photography of target lesion at select sites only
  - TLSS
- Physical Exam
- Vital Signs
- Drug dispensation / collection
- Adverse events
- Cutaneous adverse events

#### 4.2 Study Treatment

## 4.2.1 Details of Study Treatment

Enstilar® Foam is a white to off-white opalescent liquid in a pressurized aluminum spray can with a continuous valve and actuator. At administration the product is a white to off-white foam after evaporation of the propellants. Each gram of Enstilar® Foam contains 52.2 mcg calcipotriene

hydrate (equivalent to 50 mcg of calcipotriene) and 0.643 mg of betamethasone dipropionate (equivalent to 0.5 mg of betamethasone).

Enstilar® Foam contains calcipotriene hydrate and betamethasone dipropionate. It is intended for topical use only. Calcipotriene hydrate is a synthetic vitamin D3 analog. Chemically, calcipotriene hydrate is 9.10-secochola-5.7.10(19),22-tetraene-1,3,24-triol,24-cyclo-propylmonohydrate, (1a,3ß,5Z,7E,22E,24S) with the empirical formula C27H40O3,H20, a molecular weight of 430.6, Calcipotriene hydrate is a white to almost white, crystalline compound. Betamethasone dipropionate is a synthetic corticosteroid. Betamethasone dipropionate has the chemical name pregna-1,4-diene-3,20-dione-9-fluoro-11-hydroxy-16-methyl-17,21-bis(1 oxypropoxy)-(11β,16β), with the empirical formula C28H37FO7, a molecular weight of 504.6, a: Betamethasone dipropionate is a white to almost white crystalline powder. Enstilar® Foam is a white to off-white opalescent liquid in a pressurized aluminum spray can with a continuous valve and actuator. The propellants used in Enstilar® Foam are dimethyl ether and butane. At administration the product is a white to off-white foam after evaporation of the propellants. Each gram of Enstilar® Foam contains 52.2 mcg calcipotriene hydrate (equivalent to 50 mcg of calcipotriene) and 0.643 mg of betamethasone dipropionate (equivalent to 0.5 mg of betamethasone) in a base of white petrolatum, PPG-11 stearyl ether, mineral oil, all-rac-alphatocopherol, and butylhydroxytoluene.

## **Dispensation and Dosage Schedule**

A 4-week supply of study medication will be dispensed at baseline and applied daily from weeks 0 to week 4. Subjects will be instructed to apply study medication once per day per supplement II.

## 4.2.2 Treatment Assignment

All subjects who have signed an ICF will receive a 2-digit subject number, starting at 01. This subject number will be used to identify the subject throughout the study. When subjects qualify for the study, they will be randomized.

## Blinding

Study treatments will be provided to subjects in an open-label manner (the identity of the study treatment will be known by all parties.)

## 4.2.4 Supplies and Accountability

The pharmacist will inventory and acknowledge receipt of all shipments of study medication. All study medication must be kept in a locked area with access restricted to designated study personnel. The study medication must be stored in accordance with the instructions provided with the shipment. The pharmacist will also keep accurate records of the quantities of study medication dispensed and returned by each subject.

## 4.2.5 Treatment Compliance

Subject compliance to study treatment regimen will be assessed at each visit; study personnel will ask each subject whether they missed any applications of study medication since the previous visit.

# 4.3 Concomitant Medication/Treatment

Subjects must comply with the restrictions based on prohibited medications and treatments as detailed in the exclusion criteria. Other necessary therapies that will not interfere with the response

to treatment may be provided at the discretion of the Investigator. The use of any concurrent medication, prescription or over-the-counter drug, is to be recorded in the source document along with the reason the medication was taken.

#### 5 ASSESSMENTS OF EFFICACY

## 5.1 Affected Body Surface Area Assessment (BSA)

The area of body affected by psoriasis will be estimated as a percentage of the subjects total body surface area. As means to standardize measurements, the area of the subject's palm will be considered as 1% of total BSA.

5.2 Physician Global Assessment (PGA) – see attached table
The Investigator will grade the current severity of psoriasis as per PGA

#### 6 ASSESSMENTS OF SAFETY

## 6.1 Safety Assessments

Throughout the study, subjects will be monitored for signs and symptoms of adverse events. All adverse events and con meds will be recorded throughout study. An *adverse event* is any pathological or unintended change in the structure, function or chemistry of the body that occurs during the study, irrespective of causality, including any illness, injury, toxicity, sensitivity, or sudden death. The condition must either not be present pre-study or must worsen in either intensity or frequency during the study. A *serious adverse event* is any untoward medical occurrence, that, at any dose:

- results in death;
- is life-threatening;
- requires in-patient hospitalization or prolongation of existing hospitalization;
- results in persistent or significant disability/incapacity;
- is a congenital anomaly/birth defect; or
- is an important medical event.

An unexpected adverse event is any treatment-related adverse event, which is not identified in nature, severity, or frequency in current literature on the test product.

# 6.2.2 Adverse Event Reporting

All adverse events must be recorded by the Investigator into the CRF. The Investigator will be required to describe the adverse event, onset and stop date, severity, the course of action taken, i any, as well as any pertinent data necessary to allow a complete evaluation of the adverse event For serious adverse events (SAE), an additional report (SAE report) must be completed.

# 6.2.3 Follow-up and Final Reports

Subjects who have had a serious adverse event must be followed clinically until all parameters including laboratory values (if applicable), have either returned to normal or are otherwise explained If death was the outcome of the event on the initial SAE Report, a Follow-up/Final Report, including autopsy report, when performed, must be completed.



#### 7 STATISTICS

# 7.1 Sample Size Justification

This is a pilot study and a formal justification for the sample size is not provided. N = 28

## 7.2 Analyses

Statistical analyses will be conducted on an intent-to-treat population that includes all subjects who were enrolled and received study medication. Due to small sample size and exploratory nature of the study, descriptive statistics will be performed using SAS. Any additional statistical analyses will be performed as appropriate and detailed in the final report. All statistical tests will be two-sided and interpreted at a 5% significance level. Descriptive statistics (i.e., mean, standard deviation, etc.) will be provided for all continuous variables and frequencies for all categorical variables collected in this study. Summary tables will be used to present patient population characteristics at Baseline; data from the study questionnaires will be included. Analyses of study treatment will be performed using an ANCOVA technique with the Baseline value as the covariate provided the necessary assumptions for parametric tests are satisfied. The Wilcoxon Rank-Sum test will be used if the necessary assumptions for parametric tests are not satisfied. Mean scores will also be analyzed. Safety analyses will be performed in terms of incidence and severity of local tolerance signs and symptoms and adverse and/or unexpected events.

## 8 RESPONSIBILITIES OF THE INVESTIGATOR

#### 8.1 Good Clinical Practice

Investigators must adhere to the procedures outlined in this Study Protocol. The procedures set out in this study protocol, pertaining to the conduct, evaluation, and documentation of this study, are designed to ensure that the Investigator abides by GCP as described in the ICH Guidelines Topic E6: "Guideline for Good Clinical Practice." Compliance with these regulations also constitutes compliance with the ethical principles described in the current revision of the Declaration of Helsinki. The study will also be carried out in keeping with local legal and regulatory requirements.

#### 8.2 Ethics

The appropriate IRB must review the Study Protocol and Informed Consent Form prior to initiating the study. Any significant modifications to the IRB-approved protocol or informed consent must be made in consultation with the IRB.

# 8.3 Confidentiality of Subjects

Any information that identifies subjects with respect to this research study will be kept confidential. However, records identifying the subject may be inspected by representatives of the IRB and/or the FDA. Subjects' identity will remain strictly confidential during all record reviews, as well as in any publication that may result from this research. Subjects will be identified by study code only; their names will not be used.

## 8.4 Informed Consent

Informed consent is a process that is initiated prior to the individual's agreeing to participate in the study and continuing throughout the individual's study participation. Appropriate discussion of risks and possible benefits of this therapy will be provided to the subjects. Consent forms describing in

detail the study interventions/products, study procedures and risks will be given to the subject and written documentation of informed consent is required prior to starting intervention/administration study product.

Consent forms will be IRB approved and the subject will be asked to read and review the document. Upon reviewing the document, the investigator will explain the research study to the subject and answer any questions that may arise. The subjects will sign the informed consent document prior to any procedures being done specifically for the study. The subjects should have the opportunity to discuss the study with their surrogates or think about it prior to agreeing to participate. The subjects may withdraw consent at any time throughout the course of the trial. A copy of the informed consent document will be given to the subjects for their records. The rights and welfare of the subjects will be protected by emphasizing to them that the quality of their medical care will not be adversely affected if they decline to participate in this study.

## 8.5 Data Handling and Record Keeping

Investigators must ensure that proper source documentation for all study activities are diligently maintained and securely kept. Investigators will transfer all relevant data from source documents to the Case Report Form as stipulated in this Study Protocol and his/her signature on the Case Report Form guarantees completeness and integrity of these data. Investigators will maintain reliable study device dispensing/dosing records and will store study supplies in a secure, locked location. In addition, Investigators will ensure that all study-related source documentation and Case Report Forms will be maintained for a period of two years after the conclusion of the study.

#### 8.6 Direct Access to Source Data/Documents

Investigators must ensure that the Informed Consent Form clearly permit study-related monitoring, audits, IRB review, and regulatory inspections providing direct access to source data and documents.

# Physicians Global Assessment Psoriasis O. Clear: no signs of psoriasis (Hyper/hypopigmentation changes alone are acceptable). Plaque elevation = 0. Scaling = 0. Erythema = +/- (hyperpigmentation, pigmented macules,

diffuse faint pink or red coloration).

- \_\_\_\_1. Almost Clear: Plaque elevation = +/- (possible but difficult to ascertain whether there is slight elevation above normal skin). Scaling = +/- (surface dryness with some white discoloration). Erythema = up to moderate (up to definite red coloration).
- 2. Mild: Plaque elevation = slight (slight but definite elevation, typically edges are indistinct or sloped). Scaling = fine (fine scale partially or mostly covering lesions). Erythema = up to moderate (up to definite red coloration).
- \_\_\_\_ 3. Moderate: Plaque elevation = moderate (moderate elevation with rough or sloped edges). Scaling = coarse (coarse scale covering most or all of the lesions). Erythema = moderate (definite red coloration).
- 4.Severe: Plaque elevation = marked (marked elevation typically with hard or sharp edges). Scaling = coarse (coarse, nontenacious scale predominates, covering most of all lesions). Erythema = severe (very bright red coloration).
- 5. Very Severe: Plaque elevation = very marked (very marked elevation typically with hard, sharp edges). Scaling = very coarse (coarse, thick, tenacious scale over most of all lesions; rough surface). Erythema = very severe (extreme red coloration; dusky to deep red coloration).

## **Washout for Psoriasis Medications**

- a. Topical immunomodulators, topical vitamin D derivatives, tar, salicylic acid, anthralin or any other topical treatment for psoriasis except topical corticosteroids that they are already using within 2 weeks of baseline.
- b. Use of any biologics within 3 months baseline
- c. Use of other systemic psoriasis treatments (ie, oral retinoids, methotrexate, cyclosporine, or other immunomodulators) within 4 weeks of baseline.
- d. Use of UVB or PUVA within 2 weeks of baseline.
- e. Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half lives, if known (whichever is longer)

## **PSORIATIC BODY SURFACE AREA**

| BODY AREA | % of BODY AREA<br>AFFECTED | % of TOTAL BODY<br>SURFACE AREA | % of TOTAL BODY<br>SURFACE<br>AFFECTED |
|---|---|---|---|
| HEAD | | 10% | |
| TRUNK | | 30% | |
| UPPER LIMBS | | 20% | |
| LOWER LIMBS | | 40% | |
| TOTAL | | 100% | |

(Multiply the numerical percent of the body part affected x the % of the total body surface area for each body area. Then add the % of total body surface affected for each area to determine the total BSA. For example: If the % of the head affected is 10, multiply ten by the % of total body surface area (10% = 0.1) for a total of 1% of Total Body Surface Area.)

# PHYSICIAN EVALUATION OF TARGET PSORIASIS LESION

| Mark location of target plaque loca | ation and size: |
|---|---|
| Erythema | |
| Induration | |
| Scaling | |
| | Sum of scores |
| Definition: | |
| <b>Erythema</b> : $0 = \text{no evidence of eryt}$ | thema |
| 2 = pink coloration | |
| 4 = red coloration | |
| 6 = very red coloration | |
| 8 = extreme red colorat | tion |
| Induration: 0 = no evidence of pla | ague above normal skin level |
| | vation, above the normal skin level |
| 4 = Moderate elevatio | on with rounded or sloped edges to plaque |
| 6 = Marked elevation | with hard sharp edges to plaque |
| | ation with very hard sharp edges to plaque |
| | 1 5 1 1 |
| Scaling: 0 = No evidence of scaling | g on the legion |
| 2 = Mild mainly fine scale | es some lesion at least partially covered |
| 4 = Moderate somewhat of | oarser scale most lesion at least partially covered |
| 6 = Severe coarse thick see | ales virtually all lesion covered rough surface |
| 8 = Very severe coarse ver | ry thick scales all lesion covered rough surface |

## **ENSTILAR PATIENT INSTRUCTIONS**

Instruct patients to shake can prior to using Enstilar® Foam and to wash their hands after applying the product. Apply Enstilar® Foam to affected areas once daily for 4 weeks. Rub in Enstilar® Foam gently. Discontinue use when control is achieved. Instruct patients not to use more than 60 g every 4 days. Enstilar® Foam should not be used with occlusive dressings unless directed by a physician. Enstilar® Foam is not for oral, ophthalmic, or intravaginal use. Avoid use on the face, groin, or axillae, or if skin atrophy is present at the treatment site